CLINICAL TRIAL: NCT05209113
Title: Development and Evaluation of the Self-management Module in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Cansu Goncuoglu, Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA-20003
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
Keywords: self management; disease modifying treatments; clinical pharmacist; treatment adherence
MeSH Terms: conditions — Multiple Sclerosis; Treatment Adherence and Compliance | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial. Patient groups were determined by a biostatistician using the block randomization method. The block width is taken as 4 and seed number fixed at 123.
Who Masked: Participant
Masking Description: The patients included in the study do not know which group they will be included in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The self-management module, which will be applied only to the study group, includes the clinical pharmacist informing the patient verbally and in writing about MS disease, the importance of drug compliance, and monitoring of disease symptoms. The first interview will end after the Patient Health Engagement-PHE-s, Multiple Sclerosis Self-Management Revised-MSSM-R, Patient Assessment of Chronic Illness Care-PACIC scales and self-management module are applied to the study group by the clinical pharmacist. When the patients come to the outpatient clinic examination 4 and 8 months after the first interview, second and third face-to-face interview will be held with the clinical pharmacist and all scales will be applied again. During the second and third interview, no written and/or verbal information will be given to the patient again.
  Interventions: Other: Education
- Control Group (No Intervention): Patient Health Engagement (PHE-s), Multiple Sclerosis Self-Management Revised (MSSM-R), Patient Assessment of Chronic Illness Care (PACIC) scales will be administered to the control group patients whose medications and demographic information were obtained in the first face-to-face interview. The same scales will be repeated at the 4th month and 8th month, the self-management module will not be applied to the control group, and within this scope, the patients will not be informed by the clinical pharmacist, and the patient's routine outpatient services will continue.

INTERVENTIONS:
Other: Education — A self-management module was applied to the study group. This module includes informing the patient verbally and in writing about MS disease, the importance of drug compliance, and monitoring of disease symptoms.
  Arms: Study Group

SUMMARY:
Compared with other chronic disease states, MS patients feel more uncertainty and less control over illness and non-illness aspects of life, and as a result, they have poor self-management abilities. It was thought that providing evidence-based information and using balanced information in terms of risk/benefit in patient education would affect the patient's self management. It is thought that a developed comprehensive self-management module by clinical pharmacist will contribute to the literature and clinical practice, and will positively affect the treatment process of patients.

This study is aimed to improve the self-management of MS patients by informing them about the disease, treatment options, and appropriate drug use by the clinical pharmacist, and to analyze the effect of the self-management module in the short and long term by examining the change in patients' self-management, participation in the treatment process and care satisfaction and compliance.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, progressive central nervous system disease that cannot be cured in the light of current information. Disability, weakness, tremors, balance and movement problems, fatigue and depression are observed in the vast majority of MS patients. Compared with other chronic disease states, MS patients feel more uncertainty and less control over illness and non-illness aspects of life, and as a result, they have poor self-management abilities. Self-management can be defined as an individual's ability to manage symptoms, treatment, physical and psychological consequences of illness, and making lifestyle changes specific to living with a chronic condition. In studies, it was thought that providing evidence-based information and using balanced information in terms of risk/benefit in patient education would affect the patient's participation in the shared decision-making process. Self-management programs for MS patients are insufficient and this is a factor in the failure of self-management to be fully adopted. It was revealed that self-efficacy, perception of treatment control, and realistic MS process knowledge were associated with self-management in MS patients. It is thought that a developed comprehensive self-management module will contribute to the literature and clinical practice, and will positively affect the treatment process of patients. Clinical pharmacy is defined by the American College of Clinical Pharmacy as a health science offered by the pharmacist in order to organize the patient's drug therapy in the most appropriate way and to protect health, ensure healing and prevent disease. Accordingly, the clinical pharmacist is responsible for identifying and preventing the patient's possible problems with drug therapy (such as drug dose/dosing frequency/administration route suitability, drug interactions, side effects, compliance, education and information needs, therapeutic drug monitoring requirement), and other healthcare professionals. It takes part in cooperation with the multidisciplinary team, provides necessary information about drugs and ensures the continuation of rational drug treatment. Studies have reported that as a result of the integration of the clinical pharmacist into the MS outpatient clinic, patients' access to drugs is facilitated, care coordination and patient outcomes are improved. In addition, it has been shown that the presence of a clinical pharmacist in a multidisciplinary team contributes to increasing compliance, making drug follow-ups of patients, and improving communication with physicians. As a result of all these, the self-confidence of the patient, who played a key role in the joint decision-making model, increased and it was observed that the patients were more willing to be involved in the joint decision-making process.

The aim of this study is to improve the self-management of MS patients by informing them about the disease, treatment options, and appropriate drug use by the clinical pharmacist, and to analyze the effect of the self-management module in the short term (4 months) and long term (8 months) by examining the change in patients' self-management, participation in the treatment process and care satisfaction and compliance.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* Diagnosed with MS and using medication for at least 45 days,
* Approved by the physician to participate in the study,
* Giving written consent,
* Patients who have been in a stable disease period (attack free period) for at least 30 days

Exclusion Criteria:

* Has a disability that prevents communication,
* Involved in another clinical and/or drug trial,
* Patients who are pregnant / planning pregnancy during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Changes in the self-management scale (Multiple Sclerosis Self Management Revised) scores of patients after the implementation of the self-management module | 20 months
  Changes in patients' self-management in the short (4 months) and long (8 months) term will be evaluated using the MSSM-R scale.

SECONDARY OUTCOMES:
Changes in the patient engagement (Patient Health Engagement Scale) scores of patients after the implementation of the self-management module | 20 months
  Changes in patients' health engagement score in the short (4 months) and long (8 months) term will be evaluated using the PHE scale.
Changes in the perception of care (Patient Assessment of Chronic Illness Care-PACIC) scores of patients after the implementation of the self-management module | 20 months
  Changes in patients' perception of care in the short (4 months) and long (8 months) term will be evaluated using the Patient Assessment of Chronic Illness Care-PACIC scale.

CONTACTS AND LOCATIONS:
Overall Officials: Asli Tuncer, Study Chair — Hacettepe University Department of Neurology
Locations (1):
- Hacettepe University, Ankara, Sihhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No